CLINICAL TRIAL: NCT03787615
Title: Feasibility of Using sipIT Tools to Increase Compliance With Fluid Consumption Guidelines in Urolithiasis -Prone Subjects
Brief Title: Feasibility of Using sipIT Tools to Increase Compliance With Fluid Consumption Guidelines in Urolithiasis-Prone Subjects
Acronym: sipIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David E Conroy, Professor of Kinesiology and Human Development & Family Studies, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00010778; UL1TR002014 (NIH)
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Results first posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Urolithiasis
Keywords: kidney
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Intervention Model Description: A variety of technologies (e.g., wrist-worn sensors, smart water bottles, mobile applications) can be utilized to engage participants over time and support compliance with increasing fluid consumption.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- The sipIT tools (Other): The wrist-worn sensors used to detect a drinking event (FitBit Versa with custom algorithm), an H2OPal connected water bottle and fluid consumption monitoring mobile applications.
  Interventions: Device: sipIT tools

INTERVENTIONS:
Device: sipIT tools — Just in time drinking detection tools to promote increase fluid consumption

SUMMARY:
The purpose of this study is to examine the feasibility of using sipIT tools (i.e., wrist-worn sensors, smart water bottles, mobile applications) to increase compliance with physician-recommended fluid consumption guidelines in participants with a history of urolithiasis. The study aims to: 1) deliver notifications regarding fluid consumption to the FitBit Versa and the participant's smartphone based on the participant's assessed fluid intake, and 2) determine the acceptability of using the sipIT tools to increase fluid consumption. It is hypothesized that receiving notifications regarding fluid consumption will lead to an increased compliance in attaining fluid consumption guidelines. Further, it is hypothesized that the frequency of notifications will diminish across the study duration.

DETAILED DESCRIPTION:
Complying with fluid consumption guidelines provides a variety of health benefits. Patients with a history of urolithiasis are a segment of the population that can benefit from meeting physician-recommended fluid consumption guidelines. Preliminary studies with this population have revealed patient interest in using various technologies (i.e., wrist-worn sensors, smart water bottles, mobile applications) to increase their fluid consumption but the investigators are not aware of any that combine multiple technologies. The investigators' long-term goal is to examine if just-in-time reminder notifications to drink following periods when patients have not been drinking will increase compliance among patients with a history of urolithiasis. To prepare for that study, the investigators seek to evaluate the feasibility and acceptability of the sipIT tools in this study.

This study is part three of a set of studies aimed at determining the feasibility of using technology to increase compliance with fluid consumption guidelines. Preliminary data included 1) a focus group of participants with a history of urolithiasis and 2) a lab study to examine the feasibility of using wrist-worn sensors to detect non-alcoholic drinking events. Data from the focus group revealed that participants are interested in using a variety of technologies (e.g., wrist-worn sensors, smart water bottles, mobile applications) to assist with increasing fluid consumption. Data from the lab study revealed that using wrist-worn inertial sensors to detect drinking events is feasible. Based on data from the lab study, an algorithm was developed to detect these drinking events and has been implemented in a consumer smartwatch consumer smartwatch app for just-in-time drinking detection.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in spoken and written English, and capable of providing informed consent
* Own an iPhone (version 6 or higher)
* History of urolithiasis
* Willingness to complete all study procedures: completing questionnaires, participating in semi-structured interviews, tracking fluid consumption, wearing a FitBit Versa and receiving notifications on the FitBit and their smartphone for a three-month period

Exclusion Criteria:

* Any medical condition that interferes with regular fluid consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Conroy, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data with other researchers.

REFERENCES:
- [Derived] Conroy DE, West AB, Brunke-Reese D, Thomaz E, Streeper NM. Just-in-time adaptive intervention to promote fluid consumption in patients with kidney stones. Health Psychol. 2020 Dec;39(12):1062-1069. doi: 10.1037/hea0001032. PMID 33252930

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The sipIT Tools
Started | 31
Completed | 27
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | The sipIT Tools
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Intervention Assessed by Study Completion
Description: Participants who continue to use the sipIT tools (app, connected water bottle, and smartwatch) at 3 month follow-up
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | The sipIT Tools
Number analyzed (Participants) | 31
Participants | 27

2. Secondary Outcome: Difficulty of Use Subscale of the User Burden Scale
Description: Difficulty of Use subscale of the User Burden Scale (Suh et al., 2016).
Time Frame: 3 months
Population: Completers at 3-months only
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- sipIT Group Completers @ 3 Months: Participants who completed 3-month follow-up
Arm/Group | sipIT Group Completers @ 3 Months
Number analyzed (Participants) | 27
score on a scale | NA (NA) — In analyses, we found that six items had no variance and all items had mean values <1. Because of these skewed distributions and the restricted range indicative of little to no user burden, most sub-scale internal consistency estimates were not acceptable so scores from this measure were not calculated.

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | The sipIT Tools
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT03787615/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT03787615/ICF_002.pdf